CLINICAL TRIAL: NCT06868420
Title: Efficacy of Play Therapy for the Reduction of Perioperative Anxiety in Pediatric Patients Aged 3 to 6 Years Undergoing Inguinal Hernioplasty
Brief Title: Efficacy of Play Therapy for the Reduction of Perioperative Anxiety in Pediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Guadalajara (Other)
Responsible Party: Principal Investigator, ERIKA MARTINEZ-LOPEZ, PhD, Principal investigator, University of Guadalajara
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PL4Y-2024
Record Dates: First submitted 2025-02-19; First posted 2025-03-11 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2024-04

CONDITIONS: Perioperative Anxiety
Keywords: Pediatric Surgery; Anxiety Assessment; Herniorrhaphy; Play Therapy; Perioperative Anxiety
MeSH Terms: interventions — Play Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CONTROL / STANDARD CARE (No Intervention): This group received standard care, including oral midazolam (0.1 mg/kg) as an anxiolytic before surgery.
- Play Therapy With Transport Cart (Experimental): This group received a play-based intervention consisting of five minutes of play with a toy transport cart, after which the child was transported to the operating room using the same cart.
  Interventions: Behavioral: Play therapy with transport cart

INTERVENTIONS:
Behavioral: Play therapy with transport cart — he intervention consisted of allowing pediatric patients to engage in five minutes of play with a toy transport cart, after which they were transported to the operating room in the same cart.
  Arms: Play Therapy With Transport Cart

SUMMARY:
The goal of this randomized controlled clinical trial was to determine the efficacy of play therapy in reducing perioperative anxiety in pediatric patients aged 3 to 6 years undergoing inguinal hernia surgery.

The main research question was:

Was play therapy effective in reducing perioperative anxiety levels in pediatric patients undergoing inguinal hernia repair?

Primary outcome measure: Anxiety level.

Patients were randomized into two groups:

1. an intervention group, which received play therapy involving a transport cart and toys; and
2. a control group, which received anxiolytic medication and standard care.

Researchers compared the control group and the play therapy group to evaluate differences in anxiety levels using the Visual Analog Scale for Parents (VAS-P) and the Modified Yale Preoperative Anxiety Scale-Short Form (mYPAS-SF).

DETAILED DESCRIPTION:
Design and Study Population:

A randomized controlled clinical trial with parallel groups was conducted involving pediatric patients aged 3 to 6 years who were scheduled for inguinal hernia repair at Dr. Juan I. Menchaca Civil Hospital in Guadalajara, Mexico. Participants were randomly assigned to one of two groups: the play therapy group or the control group.

The play therapy group received a play-based intervention using toys. After five minutes of playing with a transport cart, the children were transported to the operating room in the same cart.

The control group received oral midazolam (0.1 mg/kg). After five minutes, they were transferred to the operating room either in a caregiver's arms or on a standard stretcher.

The study was approved by the Ethics and Research Committees (60/HCJIM-JAL/2023).

Assessment and Management of Anxiety:

Perioperative anxiety was assessed using two instruments:

The Modified Yale Preoperative Anxiety Scale-Short Form (mYPAS-SF), completed by the anesthesiologist.

The Visual Analog Scale for Parents (VAS-P), which measured anxiety as perceived by the child's parent or guardian.Both instruments were applied at three time points:

1. Upon initial contact with the anesthesiologist
2. After the intervention (play-based or pharmacological)
3. Upon arrival in the operating room Additionally, midazolam was administered as rescue therapy for any patient exhibiting significant anxiety (mYPAS-SF score > 30 following the intervention).

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients aged 3 to 6 years.
* Patients of any sex.
* Patients scheduled for elective inguinal hernioplasty.
* Patients undergoing their first anesthetic-surgical procedure.
* Patients whose legal guardian provided informed consent.

Exclusion Criteria:

* Patients with known allergy to midazolam.
* Patients with abnormal perinatal history (e.g., neonatal hypoxia or chromosomal abnormalities).
* Patients undergoing emergency inguinal hernioplasty due to complications such as strangulation or incarceration.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2023-01-19 (Actual); Primary Completion 2023-07-23 (Actual); Study Completion 2024-03-20 (Actual)

PRIMARY OUTCOMES:
Parental Assessment of Child Anxiety Levels | Baseline (pre-intervention), 5 minutes after the intervention (post-intervention), and 1 hour after the intervention (final assessment).
  The child's anxiety levels were assessed by their parent or legal guardian using the Visual Analog Anxiety Scale for Parents (VAS-P). Baseline anxiety was measured at the first contact with the anesthesiologist. The VAS-P is a 10 cm horizontal scale, where values greater than 5 cm indicate significant anxiety.
Anesthesiologist Assessment of Child Anxiety Levels | Baseline (pre-intervention), 5 minutes after the intervention (post-intervention), and 1 hour after the intervention (final assessment).
  The child's anxiety levels were assessed by the anesthesiologist using the Modified Yale Preoperative Anxiety Scale-Short Form (mYPAS-SF). Baseline anxiety was recorded at the first contact with the anesthesiologist. The mYPAS-SF provides scores ranging from 22.9 to 100 points, with values greater than 30 indicating the presence of significant anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Guadalajara, Guadalajara, Jalisco, Mexico